CLINICAL TRIAL: NCT06570239
Title: Efficacy of Spa Management (Hydrokinesitherapy and Crenobalneotherapy) Compared With Usual Management of People With Post-Covid-19 Conditions: a Randomized, Open-label Clinical Trial.
Brief Title: Evaluation of the Effectiveness of a Spa Treatment for People With Post-Covid 19 Conditions.
Acronym: COVIDTHERM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, KANNY Gisele, Professor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021PI165; 2023-A01261-44 (Other: ID-RCB)
Record Dates: First submitted 2024-07-23; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Post COVID-19 Condition

STUDY DESIGN:
Intervention Model Description: This is a regional multicentre randomised controlled open-label study. Control arm : dry support and rehabilitation protocol for 3 weeks Intervention arm: support and rehabilitation protocol in natural mineral water for for 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol A: Control group (Active Comparator): Protocol A combines dry physiotherapy with psychological support. psychological support.
  Interventions: Procedure: intervention group
- Protocol B: Intervention group (Experimental): Protocol B combines hydrokinesitherapy and hydrothermal treatments, psychological psychological support.
  Interventions: Procedure: intervention group

INTERVENTIONS:
Procedure: intervention group — Protocol A combines dry physiotherapy and psychological support. It will be organised on an outpatient basis. Weeks 1, 2 and 3: 8 sessions of "dry" physiotherapy and 3 sessions of psychotherapy. 5 psychotherapy sessions will be given over the following five weeks.
  Protocol B combines hydro-physiotherapy and hydro-thermal treatments with psychological support. Protocol B begins with 3 weeks in a spa establishment - Care provided during weeks 1, 2 and 3: 8 hydrokinesitherapy sessions, 32 hydrothermal treatments, 3 psychotherapy sessions. 5 psychology sessions will be given over the following five weeks.

SUMMARY:
Following the acute phase of Covid-19, some patients experience persistent or recurrent symptoms. These symptoms can take a number of forms: intense fatigue, cognitive dysfunction, respiratory difficulties, maladaptation to physical exertion, musculoskeletal pain, anxiety-depressive disorders, malnutrition, loss of sense of smell, headaches and so on. These symptoms are known as post-covid-19 disease, defined by the WHO as "a condition occurring in people with a history of probable or confirmed infection with SARS-CoV-2, usually 3 months after the onset of COVID-19 with symptoms that persist for at least 2 months and cannot be explained by another diagnosis. Common symptoms include fatigue, breathlessness and cognitive dysfunction, as well as other symptoms that generally have an impact on daily functioning.

The aim of this interventional research project is to assess the place of a specific spa treatment for people with a post-Covid 19 condition in the primary care pathway.

DETAILED DESCRIPTION:
Justification/context

Most of the studies initially published involved cohorts of patients hospitalized during the initial phase. The French Covid-19 cohort, which studied 1137 patients after hospitalization for SARS-CoV-2 infection, showed that 60% complained of at least one symptom still present at 6 months, 24% three or more persistent symptoms, and that 29% of those with a professional activity had not returned to work (1). At 12 months, 34% of women and 23% of men were still on sick leave (2). The susceptibility of adults seems to increase with age, number of symptoms in the acute phase, body mass index, female sex and absence of vaccination (3). The evolution of post-covid disease fluctuates over time (4).

Studies of cohorts of patients followed up in primary care show that post-covid affliction affects people with both severe and mild forms of the disease. As part of the virtual ambulatory follow-up program (CoviCare), 410 people testing positive for COVID-19 at Geneva University Hospital were followed up 7 to 9 months after diagnosis: 39.0% reported residual symptoms. Analysis of a prospective cohort of 247 Norwegian patients followed at home showed that 52% of young adults aged 16 to 30 had symptoms at 6 months, including loss of taste and/or smell (28%), fatigue (21%), dyspnea (13%), impaired concentration (13%) and memory impairment (11) A literature review of quality of life in post-covid conditions conducted between March 2020 and March 2021 (12 studies involving 4828 patients) showed that the combined prevalence of poor quality of life (EQ-VAS) was estimated at 59%. Meta-regression analysis showed that poor quality of life was significantly higher in patients with ICU admission and fatigue. At 2 months, an alteration in quality of life defined by a 10-point difference on the EQ-5D-5L analog scale was noted in 44% of hospitalized patients. The study by Logues et al, involving 177 patients in the United States, showed that 30% of outpatients had an altered quality of life at 9 months, defined as a 10-point decrease in the EQ-VAS compared with the previous situation, versus 2% of non-infected control subjects. Menges et al studied quality of life using the EQ-5D-5L scale in 431 patients in Zurich, 89% of whom were non-hospitalized. They showed that 53% of participants reported difficulties in at least one dimension of the EQ-5D-5L. The dimensions most frequently affected were pain/discomfort (39%) and anxiety/depression (31%).

Primary objective:

To compare the efficacy of a spa-based rehabilitation and support protocol (Protocol B) versus a conventional primary care rehabilitation and support protocol (Protocol A) on changes in overall quality of life at 2 months in patients suffering from post-Covid-19 symptoms who did not warrant́ hospitalization for treatment of the initial phase of Covid

Secondary objectives:

The secondary objectives of this project are:

* Compare changes in overall quality of life at 12 months between Protocols A and B.
* Compare short- (M2) and medium- (M12) term changes in persistent symptoms between Protocols A and B.
* Compare short (M2) and medium (M12) term changes in other dimensions of quality of life according to Protocols A and B: mobility, autonomy, usual activities, pain/discomfort, anxiety/depression.
* Compare the effect of protocol B versus protocol A on return to work (nature, delay and volume).
* Analyze post-covid-19 symptom profiles and their association with post-infection quality-of-life trajectories.
* Analyze and compare the mechanisms and conditions of efficacy of protocols A and B (dose of intervention received, appropriateness of the intervention to the realities of the field and the needs of the target population, patient commitment and satisfaction).

Primary outcome:

The primary endpoint of this study is the change in utility score derived from quality of life and measured by the EQ-5D-5L at inclusion (V0) and at 2 months after inclusion (V2).

Secondary outcomes:

* Variation in mean utility score (EQ-5D-5L) calculated in each management group (protocol A and protocol B) between V0 and V3, V4 and V5 (including Vend).
* Variation in the following parameters : number of symptoms and symptom clusters, rating by symptom scales and tests (Appendices), asthenia (Chalder fatigue scale (5) sleep disorders (Insomnia Severity Index́ (ISI) (6)), pain (visual analog pain scale (25)), anxiety-depression (HAD scale (7), post-traumatic stress (PCL-5 scale (8)), dyspnea (mMRC-modified Medical Research Council scale) and modified Borg scale (9,10)), lower-limb muscular strength (standing-sitting test, (11,12), 6-minute stepper test (13), postural balance on posturography platform, with sensitization by modification of somato-sensory afferents (foam tray) and visual (virtual realitý goggles) (14,15), balance tests (monopodal support eyes open and closed).
* Variation in scores for the 5 items and the visual analog scale (VAS) comprising the EQ-5D-5L questionnaire.
* Data on return to work (time taken to return to work part-time or full-time, modified post, etc.).
* Number of medical consultations, consumption of physiotherapy, psychology and other paramedical care, analgesics, anxiolytics, antidepressants, systemic or inhaled corticoids, bronchodilators and antihistamines not included in the protocol.

Methods:

This is a regional multicenter randomized controlled open-label study. Patients will be randomized 1:1 per center into two different intervention arms:

* Control arm (Protocol A): dry rehabilitation protocol for 3 weeks and psychological support for 8 weeks
* Intervention arm (Protocol B): natural mineral water rehabilitation protocol for 3 weeks and psychological support for 8 weeks.

Each included patient will be followed-up for one year with 5 different visits: at inclusion (V0), at one month (V1), at 2 months (V2), at 6 months (V3) and at 12 months (V4).

Number of research participants required:

Randomization will be 1:1 per center, and the primary endpoint is the utility score derived from quality of life and measured by the EQ-5D-5L ranging from 0 (state corresponding to death) to 1 (state of perfect health). We set an alpha risk of 5% and a power of 80%. Estimating a standard deviation of the utility score between the two groups of 0.12 and a minimum difference to be highlighted of 0.05 (equivalent to 5 points out of 100), we will need to include 91 patients per group, for a total of 182 patients. Assuming 10% drop-out during the treatment period (first 3 weeks), we need to include a total of 200 patients in the 4 selected spa centers (Amnéville, Contrexéville, Vittel and Nancy).

Inclusion capacity in the various centers is as follows: Amnéville (60), Contrexéville (30), Vittel (30) and Nancy (80).

Inclusion criteria for research subjects

* Patients who have received full information on the organization of the research, who have not objected to their participation and to the use of their data, and who have given their free and informed consent in writing,
* Patients aged 18 and over,
* Patients with a history of symptomatic Covid-19 infection documented by RT-PCR, antigenic test, positive serology in a previously unvaccinated patient or other validated virological diagnostic test at the patient's inclusion date,
* No hospitalization for treatment of the initial phase of Covid-19,
* Person presenting at least two common symptoms of post-Covid disease, including fatigue, shortness of breath and cognitive dysfunction, which have appeared de novo and have been evolving for more than 12 weeks and present for more than 8 weeks,
* Initial and prolonged symptoms not explained by another diagnosis with no known link to Covid-19,
* Normal SpO2 at rest not decreasing beyond 4% on exercise,
* Membership of a social security scheme or beneficiary of such a scheme

Criteria for non-inclusion of research subjects:

* Acute cardiovascular disease (acute coronary syndrome, arrhythmia, heart failure, venous thromboembolism, myocarditis, stroke, acute ischemia, etc.) less than 3 months old and at risk of recurrence or decompensation,
* Respiratory disease: COPD, interstitial fibrosis, exercise-induced desaturation, sleep apnea,
* Stroke less than 6 months old,
* Pregnant women,
* adults under legal protection (guardianship, curatorship, safeguard of justice),
* Severe and unstabilized psychiatric pathology, severe depressive syndrome, delirious decompensation, panic attacks, anxiety-depression syndrome,
* Acute and progressive conditions (infectious, cancerous and inflammatory),
* Persons presenting a contraindication to hydrokinesitherapy and crenotherapy (infected dermatoses, severe immune deficiencies, inflammatory diseases in flare-ups, fecal or urinary incontinence, presence of a suprapubic or intravenous catheter, colostomy, hydrophobia.
* Refusal to sign the free and informed consent form

Recruitment of research subjects (patients, controls where applicable):

The pre-selection of patients will be carried out by the structures dedicated to the care of patients suffering from post-covid conditions in the region: general practitioners, infectious disease specialists, physical medicine and rehabilitation specialists, physiotherapists. They will present the project and hand out the newsletter.

Are specially protected persons concerned? no

Prohibited period:

The person must not be included in any other intervention research during the treatment period for this research. The blackout period corresponds to the period between the inclusion visit at V0 and the V2 visit carried out at the end of the treatment period (2 months after the inclusion visit).

Compensation No compensation is planned for participants in the COVIDTHERM study.

Duration:

The inclusion period is scheduled to last 12 months, and each patient will be followed up for 12 months, for a total of 24 months

Investigation procedures and differences from usual care:

General principle:

Physiotherapists will be trained to harmonize their practices and adapt them to the specific situations of patients with post-Covid symptoms. Psychotherapy sessions will be carried out via teleconsultation, with the aim of facilitating and harmonizing the care of patients included in the study, regardless of their place of residence. Health education materials will be given to patients at the start of the treatment period, when the first assessment is carried out. Topics covered will include Understanding the post-covid condition; Understanding the psychological repercussions; Managing breathing; Managing effort; Rehabilitating the sense of smell; Managing stress; Adapting diet.

For both arms of the study, specific procedures include 3 visits to the study's investigating physician, 5 physiotherapy check-ups and 1 psychological check-up. Participants will be recruited from the population living near the resorts. Transport costs will be covered as part of the study. The prospective resorts in the Grand Est region are : Nancy Thermal, Amnéville-les-Thermes, Contrexéville and Vittel.

Protocol A: Control group Protocol A combines dry physiotherapy, psychological support and health education.

9 outpatient physiotherapy sessions over 3 weeks in the offices of private physiotherapists taking part in the study, or in suitable care facilities agreeing to take part.

1 initial psychological assessment followed by 7 psychological teleconsultations (1/week).

Protocol B: Intervention group Protocol B combines hydrokinesitherapy and hydrotherapy, psychological support and health education (kit containing health education materials).

9 hydrokinesitherapy sessions and 36 hydrothermal treatments* will be carried out over 3 weeks in one of the spa establishments participating in the study and close to the patient's place of residence.

*Hydrothermal treatments include affusion massage, jet shower, aerobath and pool mobilization, corresponding to 4 treatments three times a week for 3 weeks.

Group A and B patients will receive psychological support over an 8-week period. This will include an assessment and 7 teleconsultations (1/week).

Acts requiring logistics :

* Training of Covid Long staff (doctors, physiotherapists).
* Patient questionnaires.
* Organization of psychology teleconsultations.
* Organization of semi-structured interviews

Nature and origin of the data collected:

Type of data collected for the study :

Sex - age Socio-professional category Family status Health data Covid-19 health data Lifestyle and behavior Working life Lifestyle Location Autonomy Physical abilities Activities of daily living Breathing capacity Neurological disorders Motor functions and musculoskeletal capacities, upper and lower limbs and spine Medical data will be collected from the medical records of the investigating physicians. Socio-demographic and perceived health data will be collected via self-administered questionnaires administered administered to patients. Individual semi-structured interviews will also be conducted with professionals and a sub-sample of 10% of patients, i.e. 20 patients randomly selected and having indicated that they would be willing to participate in an interview conducted at the end of the interventions (M2).

Method of collecting personal data:

The clinical, sociodemographic and perceived health data collected will be entered on an electronic CRF, then stored on a secure server at the CHRU de Nancy in accordance with quality procedures.

Circulation of personal data and procedures for protecting confidentiality:

An anonymity number will be created for each patient. This number will be made up of 4 digits, the first corresponding to the center number and the next three to the number assigned at inclusion in chronological order. The first patient in center 1 will have the number 1 001, and the first patient in center 4 will have the number 4 001.

A correspondence table will be kept securely at each investigating center to link the study number to the subject's identity.

Assessing the benefits and risks of research:

Expected benefits

* Validation of the effectiveness of rehabilitative and supportive care in the management of people suffering from post-covid symptoms,
* Demonstration of the superiority of hydrokinesitherapy and crenotherapy over conventional rehabilitation in primary care, with both protocols performed in accordance with HAS recommendations,
* Validation of a specific care pathway adapted to patients with persistent symptoms following Covid-19.
* Provision of a dedicated care pathway for primary care physicians, with health professionals trained and available for this type of care.

The risks are those associated with :

* dry rehabilitation: risk of over-intensive rehabilitation
* hydrokinesitherapy rehabilitation: risk associated with thermoregulation disorders in an aquatic environment
* thermal treatment
* infections transmitted by other spa guests (mainly benign ENT infections)
* legionellosis: risk controlled by hygiene measures introduced in spa establishments (decree of June 19, 2000 on the management of microbial risk linked to mineral water in spa establishments),
* Risk of slips and falls in the establishment.

Statistical analysis:

The program's primary efficacy criterion will be assessed by comparing mean changes in the overall quality of life score (utility score) at 2 months between the two groups. An analysis of missing data will be performed, and the random or non-random nature of missing data will be investigated (Diggle and Rubins classification). Two types of analysis will be used for the main analysis: a univariate analysis to compare differences in quality of life scores between the two arms: non-parametric (Mann Whitney-Wilcoxon) and/or parametric (Student's t test); a multivariate analysis of variance on repeated measures with adjustment for potential confounding variables (clinical and socio-demographic, and center). A pairwise analysis will also be used to perform a combined analysis of several judgment criteria (quality of life, anxiety, etc.) with their prioritization.

Expected benefits Reduce the intensity, duration and impact on quality of life of persistent post-Covid symptoms, and enable resumption of social and professional activities; Provide French primary care physicians with a dedicated network of healthcare professionals trained and available for this type of care; Position spa treatment within the healthcare pathway of people with post-covid conditions; Provide state-of-the-art symptom management for this emerging pathology; Better understand the natural history of post-covid symptoms.

Funding:

This project is co-financed by the following organizations:

* Agence Régionale de Santé ARS-Grand Est,
* CNETh (Conseil National des Établissements Thermaux),
* Région Grand Est,
* Metropole du Grand Nancy.

A budget of 207,000 euros has been obtained.

Research schedule and organisation:

Inclusion period: 1 year Duration of follow-up period: 1 year Overall study duration (including analyses): 30 months

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information about the organisation of the research, who has not
* to their participation and the use of their data, and who have given their free and free and informed consent in writing,
* Patients aged 18 and over,
* Patients with a history of symptomatic Covid-19 infection documented by RTPCR, antigenic test, positive serology in a patient not previously vaccinated or other virological diagnostic test validated at the patient's inclusion date,
* A person who has not required hospitalisation for treatment in the initial phase of Covid-19,
* Person presenting at least two common symptoms of the post-Covid condition from among fatigue, breathlessness, cognitive dysfunction, appearing de novo and evolving for more than for more than 12 weeks and present for more than 8 weeks,
* Initial and prolonged symptoms not explained by another diagnosis with no known link to with Covid-19,
* Normal SpO2 at rest not decreasing beyond 4% on exercise,
* Membership of a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Acute cardiovascular disease (acute coronary syndrome, arrhythmia, heart failure, venous thromboembolism venous thromboembolic disease, myocarditis, stroke, acute ischaemia, etc.) less than stroke, acute ischaemia, etc.) less than 3 months old and at risk of recurrence or decompensation,
* Respiratory disease: COPD, interstitial fibrosis, exercise-induced desaturation, sleep apnoea
* Stroke less than 6 months old,
* Pregnant women,
* Adults subject to a legal protection measure (guardianship, curatorship, safeguard of justice),
* Serious and unstable psychiatric pathology, severe depressive syndrome, delirious decompensation, panic attacks, anxiety-depression syndrome,
* Acute and progressive conditions (infectious, cancerous and inflammatory),
* Person with a contraindication to hydrokinesitherapy and crenotherapy crenotherapy (infected dermatoses, severe immune deficiencies, inflammatory diseases, faecal or urinary incontinence, presence of a suprapubic or intravenous catheter, colostomy, hydrophobia)
* Refusal to sign the free and informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | at the 2-month visit (V2)
  The primary endpoint of this study was the change in the utility score derived from the measured by the EQ-5D-5L at 2 months (V2-V0) after inclusion.

SECONDARY OUTCOMES:
Utility score (EQ-5D-5L) | Utility score (EQ-5D-5L) measured at the 2-month visit (V2), the six-month visit (V3) and the 12-month visit (V4)
  Variation in the mean utility score (EQ-5D-5L) calculated in each management group (protocol A and protocol B) between V0 and V2, V3 and V4 (including Vend),
Number of symptoms and symptoms clusters | Utility score (EQ-5D-5L) measured at the 2-month visit (V2), the six-month visit (V3) and the 12-month visit (V4)
  Variation in the following parameters: number of symptoms and symptoms clusters, scoring by symptom scales and tests (Appendices), asthenia (Chalder fatigue scale ), sleep disorders (Insomnia Severity Index́ (ISI) ), pain (visual analogue pain scale ), anxiety-depression (HAD scale ), post-traumatic stress (PCL-5 scale ), dyspnoea (mMRC - modified Medical Research Council scale) and modified Borg scale , muscle strength in the limbs (standing-sitting test ), balance tests (FUKUDA test, get up and go test), postural balance on a posturography platform, with sensitisation by modification of somato-sensory afferents (foam tray) and visual afferents (goggles virtual realitý goggles),
Return to work | Employment status requested at the 2-month visit (V2), the six-month visit (V3) and the 12-month visit (V4)
  Data on return to work (time taken to return to work part-time and full-time, modified post, etc.),
Medical consultations | Number of medical consultations at the 2-month visit (V2), the six-month visit (V3) and the 12-month visit (V4)
  Number of medical consultations, physiotherapy, psychology and other paramedical psychology and other paramedical care, analgesics, anxiolytics, anti-depressants, systemic or inhaled corticosteroids, bronchodilators and antihistamines not included in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Giséle KANNY, PU-PH, Principal Investigator — CHRU de Nancy; Julie DALCOURT, PH, Principal Investigator — Centre Hospitalier Ouest Vosgien CHOV; Simon RUDYNSKI, Dr, Principal Investigator — Centre Thermal Saint Eloy-Amnéville